CLINICAL TRIAL: NCT05356754
Title: PROSPECTIVE STUDY EVALUATING THE VITAL LABS DIGITAL BLOOD PRESSURE MONITOR (VLDBPM)
Brief Title: VL-3 Training Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riva Health (Industry)
Collaborators: Diablo Clinical Research (Unknown); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP-0001
Record Dates: First submitted 2022-04-22; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Hypertension; Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- The Vital Labs Digital Blood Pressure Monitor (Experimental): The Vital Labs Digital Blood Pressure monitor is a software-as-a-medical device (SaMD) that is capable of determining blood pressure, after calibration, using waveform changes observed in photoplethysmogram signals. The VLDBPM captures PPG signals using the existing camera systems on iPhones. These PPG signals are normalized and processed to determine markers of blood pressure change. These markers, when transformed using a predetermined model, are capable of determining blood pressure changes from a known (calibration) set-point.
  Interventions: Device: The Vital Labs Digital Blood Pressure Monitor

INTERVENTIONS:
Device: The Vital Labs Digital Blood Pressure Monitor — The Vital Labs Digital Blood Pressure monitor is a software-as-a-medical device (SaMD) that is capable of determining blood pressure, after calibration, using waveform changes observed in photoplethysmogram signals.

SUMMARY:
The primary endpoints for this study are mean and standard deviation error measurements for the VLDBPM versus manual auscultation.

DETAILED DESCRIPTION:
This is a prospective, controlled, single-arm clinical evaluation. Five hundred thirty-two (532) subjects are planned to be evaluated. Each subject's blood pressure will be measured using the VLDBPM and manual auscultation. Each subject will be observed while undergoing a series of blood pressure perturbation challenges. Means measurement differences from the test sensor and the reference auscultation measurements will be used to validate the accuracy of the VDBPM software system.

Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study.

Total duration of subject participation will be 1 to 1.5 hours. Total duration of the study is expected to be 6 months.

Following medical history and patient eligibility assessments, eligible patients will be offered participation in the study. Once subjects are consented/enrolled, measurements will be performed in accordance with Data Collection Procedure section below.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 and ≤ 85 years of age at the Baseline Visit.
* Written informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.
* A minimum of 30% of the data will be derived from male subjects; and a minimum of 30% of the data will be derived from female subjects.
* A minimum of 50 participants will have dark skin types, as defined by the Fitzpatrick Skin Type classification V or VI.
* Also, at least 10 participants should exhibit finger calluses, found typically on individuals who play stringed instruments frequently.

Exclusion Criteria:

* 1. Pregnant and/or breastfeeding. 2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

  3. Are unable or unwilling to undergo all assessments associated with the study.

  4. Have a history of poor quality or difficulty performing auscultation measurements.

  5. Subjects shall be excluded if the Korotkoff sound [fifth phase (K5)] is not audible 6. Subjects with vascular implants in the arm of measurement, such as those used for dialysis 7. Subject suffering from a medical condition prohibiting blood flow occlusion in either arms.

  8. Pre-existing conditions that may interfere with the accuracy or interpretation of auscultatory readings, such as aortic coarctation, arterial-venous malformation, occlusive arterial disease, or the presence of an antecubital bruit.

  9. Subjects who have known allergies to nitroglycerin (for subjects undergoing the nitroglycerin challenge).

  10. Subjects who have taken short acting nitroglycerin within 4 hours of the scheduled study. Such studies will be deferred for at least 4 hours.

  11. Subjects who have taken long acting nitroglycerin within 8 hours of the scheduled study. Such studies will be deferred for at least 8 hours.

  12. Subjects with pericardial tamponade, restrictive cardiomyopathy, or constrictive pericarditis, or cardiac output is dependent upon venous return

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Mean difference between BP measures | Baseline
  Primary efficacy
Standard deviation of differences between BP measures | Baseline
  Primary Efficacy
Mean difference between BP measures | 1.5 hours
  Primary efficacy
Standard deviation of differences between BP measures | 1.5 hours
  Primary Efficacy

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - Diablo Clinical Research, Walnut Creek, California
  - University of Colorado Hospital, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No